CLINICAL TRIAL: NCT05626764
Title: Monitoring Multidimensional Aspects of QUAlity of Life After Cancer ImmunoTherapy, an Open Smart Digital Platform for Personalized Prevention and Patient Management - QUALITOP -
Brief Title: QUALITOP - Monitoring Multidimensional Aspects of QUAlity of Life After Cancer ImmunoTherapy, an Open Smart Digital Platform for Personalized Prevention and Patient Management
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 346
Record Dates: First submitted 2022-10-25; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Solid Tumor; Hematologic Cancer
Keywords: hematologic tumor; immunotherapy; immune checkpoint inhibitor; CAR-T cell; cancer; QoL; HR-QoL; irAEs
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immune checkpoint inhibitors: Any immunotherapy by immune checkpoint inhibitor molecule in combination or monotherapy, associated or no with any other cancer treatment such as chemotherapy, targeted therapy, radiotherapy, etc.
  Interventions: Other: QoL & irAEs determinants
- CAR-T cells: Transplantation of recombined autologous immune T-cells
  Interventions: Other: QoL & irAEs determinants

INTERVENTIONS:
Other: QoL & irAEs determinants — Assesment of the QoL & irAEs determinants in patients diagnosed with solid tumor and treated in France, Netherlands, Portugal, Spain, with immunotherapy by immune checkpoint inhibitors.
  Groups: Immune checkpoint inhibitors
Other: QoL & irAEs determinants — Assesment of the QoL & irAEs determinants in patients diagnosed with hematologic cancer and treated in France, Netherlands, Portugal, Spain, by CAR-T cells.
  Groups: CAR-T cells

SUMMARY:
An increasing number of cancer patients are eligible to receive immunotherapy. Efficacy and tolerance have been demonstrated in multicentre randomized clinical trials with positive results. However, real-life experience differs from clinical trial results, especially regarding the management of potential adverse events. HR-QoL (Health Related Quality of Life) is one of the components of QoL (Quality of Life) in its broad acceptation and is certainly the only one usually collected in trials while little is known about QoL in cancer patients treated in the 'real-world'. QUALITOP partners intend to bring together all relevant longitudinal information present in large heterogeneous data (big data) to estimate patient QoL and find surrogate markers of QoL and its evolution. Within the QUALITOP consortium, 5 countries will collect prospective clinical and QoL data and also retrospective clinical data, and share it. This project will enable collecting, managing, sharing, modelling, processing, and exploiting big data on QoL. Furthermore, beyond the description of QoL, analytical tools (including causal inference methods and machine learning) are needed to understand the determinants of QoL and their complex relationships with irAEs (immune related Adverse Events) in a big-data context where standard statistical techniques would be limited. Artificial intelligence and causal models may be applied and developed to empower the patient, prevent adverse medical conditions, and promote QoL. The created knowledge will enable proposing guidelines for promoting better QoL.

QUALITOP aims at identifying the determinants of health status regarding immunotherapy-related adverse events (IR-AEs, such as toxicities) depending on the patient's profile in a real-world context.

The richness of QUALITOP is in the diversity of the experts who will collaborate in it. Clinicians involved in the care (thus the health status of the patients) will collaborate with psychologists and sociologists to understand and integrate complementary dimensions of QoL related to immunotherapy. Experts in pharmacovigilance and pharmacists will investigate the IR-AEs and their associations with patient behaviour and non-drug consumption. Epidemiologists, data scientists (including bioinformaticians and biostatisticians) and economists will extract information from the data and develop simulation models to produce knowledge. The project will take place in close relation with patient associations that will interact with experts to design the analyses, interpret their results, and proceed to their dissemination.

The main objective is to collect data of patients receiving immunotherapy in order to describe its impact in their quality of life.

* Create the first real-life cohort of cancer patients treated with immunotherapy within a context of multidimensional management (with data on clinical information, health-related QoL (HR-QoL), IR-AEs, drug consumption, lifestyle, and administrative data).
* Accelerate knowledge directed to different stakeholders (patients, relatives, clinicians, pharmacists, health authorities, and the general public) for a better understanding of the determinants of QoL and its optimization after immunotherapy through the development of innovative analytic tools (artificial intelligence and causal models).
* Produce policies and recommendations to improve patients QoL and participate in the implementation of the SDGs (Sustainable Development Goals) for 4P medicine (Predictive, Preventive, Personalized, Participative) in immunotherapy for cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* - Age > 18
* Patients starting an immunotherapy treatment by immune checkpoint inhibitor or CAR-T cells
* Patients receiving the QUALITOP informational note
* Patients receiving an immunotherapy treatment within a clinical trial could be eligible according to the promotor of the clinical trial' indications
* Patients in clinical trial which includes a combination of therapy with one of the drug administered in a blind manner vs placebo, can be eligible to QUALITOP provided that (i) the treatment administered in a blind manner is not the immunotherapy and (ii) the clinical trial allows concomitant participation of patients in non-interventional study
* Patients treated with immunotherapy by immune checkpoint inhibitors or CAR-T cells and recruited in the consortium clinical trials
* Patients in existing databases with a data sharing consent

Exclusion Criteria:

* Patients under 18
* Patients who received an immunotherapy treatment within 6 months before entering QUALITOP
* Pregnant women
* Patient refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: to define
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Assesment of the QoL& irAEs determinants in patients diagnosed with solid or hematologic cancer and treated in France, Netherlands, Portugal, Spain, with immunotherapy by immune checkpoint inhibitors or CAR-T cells. | Clinical data will be collected during 18 months starting from treatment initiation, or until the last patient reaches the 18 months follow-up. Clinical and biological changes occurring during the treatment will be assessed and compared to baseline. QoL
  Descriptive analysis of QoL determinants (which are there ? what are their impacts ? etc) based on collected data from the beginning of the treatment to 2 years.

CONTACTS AND LOCATIONS:
Locations (5):
- Medical Clinical Research Platform, Cancer Institute of the Hospices Civils de Lyon, Pierre-Bénite, France
- Netherlands (2):
  - Academic Medical Center Amsterdam, Amsterdam
  - University Medical Center Groningen, Amsterdam
- Instituto Português de Oncologia, Lisbon, Portugal
- Hospital Clinic de Barcelona - Consorci Institut d'Investigacions Biomediques August Pi i Sunyer, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vinke PC, Combalia M, de Bock GH, Leyrat C, Spanjaart AM, Dalle S, Gomes da Silva M, Fouda Essongue A, Rabier A, Pannard M, Jalali MS, Elgammal A, Papazoglou M, Hacid MS, Rioufol C, Kersten MJ, van Oijen MG, Suazo-Zepeda E, Malhotra A, Coquery E, Anota A, Preau M, Fauvernier M, Coz E, Puig S, Maucort-Boulch D. Monitoring multidimensional aspects of quality of life after cancer immunotherapy: protocol for the international multicentre, observational QUALITOP cohort study. BMJ Open. 2023 Apr 27;13(4):e069090. doi: 10.1136/bmjopen-2022-069090. PMID 37105689